CLINICAL TRIAL: NCT00174720
Title: A Multinational,Multicenter,Randomized,Double-Blind,Placebo-Controlled,Parallel-Group Study to Assess the Efficacy of Ciclesonide Metered-Dose Inhaler at a Daily Dose of 160 μg Administered Either in a Once-Daily in the Morning Regimen (160 μg qd AM) for 16 Weeks or in a 160 μg qd AM Regimen for 12 Weeks Preceded by a Twice-Daily Regimen (80 μg Bid) for 4 Weeks,or in an 80 μg Bid Regimen for 16 Weeks,in Adults and Adolescents With Mild to Moderate Persistent Asthma Not Treated With Steroids
Brief Title: Efficacy of Ciclesonide vs Placebo Administered as Once Daily or Twice Daily in Patients Not Treated With Inhaled Corticosteroid.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6164; XRP1526B/3031
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Asthma
Keywords: Glucocorticosteroid. Bronchospasm
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Ciclesonide (XRP1526)

SUMMARY:
To investigate the efficacy of ciclesonide MDI either as once daily or twice daily in patients with mild to moderate asthma, who have not previously been treated with an inhaled corticosteroid.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 12 years or older
* History of persistent bronchial asthma for at least 6 months
* Documented use of bronchodilators (short acting only) only or methylxanthines for at least 1 month before screening
* At screening, FEV1 60 to 90% of predicted. Reversibility of FEV1 by at least 12% post-bronchodilator
* Be able to use oral inhalers
* Non-smokers

Exclusion Criteria:

* History of life-threatening asthma
* Other pulmonary diseases
* URI within 4 weeks before screening
* Use of systemic steroids within 6 months before screening. Use of inhaled steroids within 30 days before screening. More than 2 in-patient hospitalizations or ER visits due to asthma exacerbations in the prior year before screening
* Pregnant or breast-feeding females
* Females of child-bearing potential not using adequate means of birth control
* Clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease
* Abnormal clinical laboratory parameters that would limit participation in the study or interfere with interpretation of study results
* History of drug or alcohol abuse
* Treatment with any investigational product within 30 days prior to study entry

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2005-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 16 in FEV1

SECONDARY OUTCOMES:
Symptom scores, rescue albuterol use and morning peak flow measurements

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (11):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, San José, Costa Rica
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Riga, Latvia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, San Juan, Puerto Rico
- Sanofi-Aventis Administrative Office, Moscow, Russia

REFERENCES:
- [Derived] Berger WE, Kerwin E, Bernstein DI, Pedinoff A, Bensch G, Karafilidis J. Efficacy and safety evaluation of ciclesonide in subjects with mild-to-moderate asthma not currently using inhaled corticosteroids. Allergy Asthma Proc. 2009 May-Jun;30(3):304-14. doi: 10.2500/aap.2009.30.3242. PMID 19549432